CLINICAL TRIAL: NCT03587012
Title: Brain Fitness APP for Cognitive Enhancement of People With Dementia
Brief Title: Brain Fitness APP for Cognitive Enhancement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Zahra Kazem-Moussavi, Professor, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018:029GB
Record Dates: First submitted 2018-04-11; First posted 2018-07-16 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Mild Cognitive Impairment; Alzheimer Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain fitness app (Experimental): Daily tutored sessions of brain exercises on an iPAD (in-person or remote)
  Interventions: Other: Brain fitness app
- Brain fitness app with tACS (Experimental): Daily tutored sessions of brain exercises on an iPAD combined with simultaneous transcranial alternating current stimulation (tACS)
  Interventions: Other: Brain fitness app with tACS

INTERVENTIONS:
Other: Brain fitness app — Daily tutored sessions of brain exercises on an iPAD (in-person or remote)
  Arms: Brain fitness app
Other: Brain fitness app with tACS — Daily tutored sessions of brain exercises on an iPAD with simultaneous transcranial alternating current stimulation (tACS)
  Arms: Brain fitness app with tACS

SUMMARY:
Memory and cognitive declines are associated with normal brain aging but are also precursors to dementia, in particular the so called the pandemic of the century, Alzheimer's disease. While currently there is no cure or "vaccine" against dementia, there are hopes to delay the onset of the disease by living a brain-healthy life style. The proposed research offers a novel approach to prevent dementia and age-related cognitive disorders.

We propose to use our developed brain fitness APP for the aging population with dementia. The proposed APP is based on the premise of brain plasticity, and targets the brain functions that are declining with normal aging and dementia. In a pilot study, we showed very positive effects of our custom designed brain exercises to strengthen left-right side brain connectivity in older adults when used regularly. Leveraging our previous design, we have developed an end-user product with additional features and enhanced user interface and user experience that will allow it to be used for neuro-cognitive rehabilitation by an individual without supervision The proposed APP will be tested on 30 individuals with cognitive impairment.

Additionally, participants can receive an optional electrical stimulation called transcranial alternating current stimulation. This applies an alternating current to a person's brain by two electrodes placed on the scalp. The participants, who choose this option, will receive simultaneous stimulation during the brain exercise tutored sessions. Studies have shown that simultaneous application of the electrical stimulation and cognitive exercises further enhances the cognitive function by boosting the working memory improvement. Thus, this may lead to further improvements from any potential positive effects of the brain exercises.

We anticipate the frequent use of the proposed APP will help to slow and even reverse the progression of the cognition decline in individuals with mild cognitive impairment or dementia.

DETAILED DESCRIPTION:
The research is on the frequent use of our designed APP (for iPADs) that contains a series of our recently developed brain exercises that contains a series of our recently developed brain exercises, including orientation, associative memory, word-image association, recall memory, etc. Participant can receive an optional electrical stimulation called transcranial alternating current stimulation (tACS) simultaneously during the brain exercise tutor sessions.

Each participant will have a dedicated tutor for Brain Exercises with three scheduling options:

A) 5 days/week, 2 sessions/day each 30 min) for a period of 4 weeks, B) 3 days/week, 2 sessions/day each 30 minute for a period of 8 weeks, C) Remote program, 5 days/week, 40min/day for a period of 4 weeks (this option is not available for participants receiving tACS).

ELIGIBILITY:
Inclusion Criteria:

* Age: 20+ years
* Have a score of 7≤ MoCA ≤ 25
* Being diagnosed with either mild cognitive impairment (MCI) or mild/moderate stage of Alzheimer's.
* Except the MCI/Alzheimer's diagnosis, have no known or diagnosis of major depression, bipolar disorder, schizophrenia, mood disorder, Parkinson's disease, Huntington disease, ALS, MS, and/or any other neurological disorder.
* Reading/writing fluency in English

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Wechsler Memory Scale (WMS IV) | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  This assessment has a total of 11 tests, out of which we will use its six primary tests that assess our target brain functions, comprised of 12 subtests (subsections): Logical Memory 1, Verbal Paired Associates 1, Faces 1, Family Pictures 1, Logical Memory 2, Verbal Paired Associates 2, Faces 2, Family Pictures 2, Verbal Paired Associates 2 Recognition, Logical Memory 2 Recognition, Letter-Number Sequencing and Spatial Span. They are classified into 3 major memory indexes: Immediate Memory, General Memory and Working Memory.

SECONDARY OUTCOMES:
Change in Egocentric Spatial Orientation | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  This test is one of the PI's designs that has been in use since a few years ago. It is used for detecting the onset of Alzheimer's. In this test participants sit in a customized wheelchair and by waking the wheelchair they move within a virtual cubic building to reach a particular target room. They can do this test either using the laptop screen or in its immersive version wearing a goggle (Oculus Rift 2).
Change in MONTGOMERY ASBERG DEPRESSION RATING SCALE (MADRS) | baseline, post-intervention within a week after the end of 4-week trial and a month after the second assessment
  The MADRS is a ten item rating scale for rating levels of depression. Each item is rated on a 7-point scale from 0 to 6, where 0 indicates absence of the symptom and 6 indicates extreme presence of the symptom. The time frame for the scale is the previous four weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided